CLINICAL TRIAL: NCT06316713
Title: Spanish Language Adaptation of One MORE for Chronic Pain in Latinos
Brief Title: One MORE for Chronic Pain in Latinos
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Eric Garland, Professor, University of Utah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB_00166637
Record Dates: First submitted 2024-03-08; First posted 2024-03-18 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Chronic Pain
Keywords: Mindfulness
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One MORE (Spanish Adaptation) (Experimental)
  Interventions: Behavioral: One MORE (Spanish Adaptation)
- Waitlist Control (No Intervention)

INTERVENTIONS:
Behavioral: One MORE (Spanish Adaptation) — One MORE is a 2-hour adaptation of the manualized MORE program and will be divided into two, 1-hour segments. In the first segment, participants will be introduced to mindfulness and guided though a body scan practice, which directs participants to systematically shift attention from one part of the body to the next. Participants will also be guided through a mindful pain management practice in which they will learn to deconstruct pain into sensory, emotional, cognitive, and behavioral components. The second segment will focus on managing the negative thoughts and emotion that can amplify pain with mindful reappraisal, as well as learning to focus on increasing the positive emotions that can attenuate pain with mindful savoring.
  Arms: One MORE (Spanish Adaptation)

SUMMARY:
This study will be a single-site, two-arm randomized controlled trial conducted among Spanish-speaking chronic pain patients. Chronic pain patients will be randomized by a computer-generated randomization schedule with simple random allocation (1:1) to either One MORE or a wait-list control condition (WLC). One MORE will be delivered individually either in-person or via a HIPAA compliant virtual meeting platform.

ELIGIBILITY:
Inclusion Criteria:

* Spanish-speaking
* Age 18+
* Diagnosed with a chronic pain condition
* Average pain in the previous week > or = 3
* Willingness to participate in study interventions and assessments.

Exclusion Criteria:

* Non Spanish-speaking
* Score of 10 or greater ('high risk') on the suicidality subsection of the MINI
* Psychotic episode within the last 12 months as deemed by the corresponding subsection of the MINI
* Presence of clinically unstable illness judged to interfere with treatment or study procedures
* Unable or unlikely to complete study procedures (e.g., planned major surgery, anticipated move, travel barrier)
* Communication or cognitive impairment that limits participation in treatment or study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity & Interference | Will be completed at baseline, week 2, and week 6.
  Change in pain intensity and interference from baseline through 6-week follow-up will be assessed with the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 30, with higher scores reflecting greater pain intensity/interference.

SECONDARY OUTCOMES:
Acute Pain | Will be completed immediately before and after each of the two, 1-hour sessions of the One MORE intervention.
  Change in acute pain will be measured with two individual items ("How much pain are you in, right now?", and "How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain.
Acceptability | Will be completed immediately after the second of the two, 1-hour sessions of the One MORE intervention.
  Acceptability will be measured with two individual items ("How acceptable did you find the strategies for managing your pain?") and ("How likely would you be to recommend this therapy to someone else dealing with chronic pain?") Scores range from 0 to 10, with higher scores indicating greater program acceptability.

OTHER OUTCOMES:
Pain Catastrophizing | Will be completed at baseline, week 2, and week 6.
  Change in pain catastrophizing from baseline through 6-week follow-up will be assessed with the Pain Catastrophizing Scale (4 question version). Scores range from 0 to 20, with higher scores reflecting greater pain catastrophizing.
Well-Being | Will be completed at baseline, week 2, and week 6.
  Change in well-being from baseline through 6-week follow-up will be assessed with the World Health Organization Well-Being Scale (5 question version). Scores range from 0 to 25, with higher scores indicating greater well-being.
Depression | Will be completed at baseline, week 2, and week 6.
  Change in depression from baseline through 6-week follow-up will be assessed with the Patient Health Questionnaire-2. Scores range from 0 to 6, with higher scores reflecting greater depression.
Anxiety | Will be completed at baseline, week 2, and week 6.
  Change in anxiety from baseline through 6-week follow-up will be assessed with the Generalized Anxiety Disorder 2-item. Scores range from 0 to 6, with higher scores reflecting greater anxiety.
Mindful Reappraisal of Pain Sensations | Will be completed at baseline, week 2, and week 6.
  Change in Mindful Reappraisal of Pain Sensations from baseline through 6-week follow-up will be assessed with the Mindful Reappraisal of Pain Sensations Scale. Scores range from 0 to 54, with higher scores indicating greater mindful reappraisal of pain sensations.
Trait Self-Transcendence | Will be completed at baseline, week 2, and week 6.
  Change in trait self-transcendence from baseline through 6-week follow-up will be assessed with the Nondual Awareness Dimensional Assessment - Trait Version. Scores range from 0 to 52, with higher scores reflecting greater trait self-transcendence.
Decentering | Will be completed immediately before and after each of the two, 1-hour sessions of the One MORE intervention.
  Change in decentering will be measured with the state version of the Metacognitive Processes of Decentering scale. Scores range from 0 to 10, with higher scores reflecting greater decentering.
State Self-Transcendence | Will be completed immediately before and after each of the two, 1-hour sessions of the One MORE intervention.
  Change in self-transcendent state will be measured with the Nondual Awareness Dimensional Assessment - State Version. Scores range from 0 to 10, with higher scores reflecting greater self-transcendence.
State Anxiety | Will be completed immediately before and after each of the two, 1-hour sessions of the One MORE intervention.
  Change in state anxiety will be measured with an individual item ("How anxious are you, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided